CLINICAL TRIAL: NCT07146204
Title: First in Human Evaluation of the R-Star, a Novel Robotic-assisted Percutaneous Coronary Intervention System
Brief Title: First in Human Trial of R-Star: A Novel Robotic System for Minimally Invasive Coronary Artery Procedures.
Acronym: R-STAR-FIH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Robocath (Industry)
Collaborators: Veranex Switzerland SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROB-04
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; percutaneous coronary intervention; Robotic-assisted percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study participants (Experimental): Patients with confirmed CAD, with indication for elective PCI
  Interventions: Device: Robotic-assisted percutaneous coronary intervention

INTERVENTIONS:
Device: Robotic-assisted percutaneous coronary intervention — Patients with coronary artery disease will be treated usiing the R-Star robotic system for a robotic-assisted percutaneous coronary intervention

SUMMARY:
The goal of this clinical trial is to learn if the R-Star robotic system can be used safely and effectively to perform percutaneous coronary intervention (PCI) in adults with coronary artery disease who are scheduled for an elective PCI.

The main questions it aims to answer are:

* Can PCI be completed with the robotic system without needing to switch fully to manual operation because of a technical issue or system limitation?
* Is the treated artery adequately opened without complications during the procedure?

Participants will:

* Have selection tests, including a medical exam, lab tests, ECG, and a review of their medical history.
* Undergo PCI using the R-Star robotic system, with angiography before and after the procedure.
* Have checkups before leaving the hospital and about 30 days later to monitor recovery and collect study data.

DETAILED DESCRIPTION:
the R-STAR PCI FIH study is a prospective, interventional, first-in-human, exploratory, single-arm, open-label, pre-marketing pilot study conducted at a single site.

This study is designed to evaluate the safety and performance of the R-Two system, as well as the clinical feasibility of its use under normal conditions of use, in accordance with the General Safety and Performance Requirements pertaining to clinical evaluation of the device, as per Annex I of the Medical Device Regulation MDR 2017/745 (EU).

The study includes four visits. The baseline visit is performed prior to the index procedure and includes subject screening and eligibility verification as well as the informed consent process. The procedure visit (Day 0) corresponds to the index RA-PCI performed with the R-Two System and includes peri-procedural assessments. The post-procedure/hospital discharge visit (Day +1) allows for early follow-up and safety evaluation. Finally, the 30-day post-procedure visit (Day 30 ±7) is conducted to assess clinical status and collect follow-up information.

Based on preclinical findings and prior experience with robotic-assisted PCI, the R-Two platform is expected to demonstrate high levels of technical and clinical performance and safety in the intended population. The system is designed to reduce operator radiation exposure and to improve ergonomics by enabling remote operation from a control room, thereby limiting physical strain. Clinical outcomes are anticipated to be favorable, with low complication rates and improved operator working conditions. Secondary endpoints, such as procedure duration, fluoroscopy time, and contrast agent volume, are also expected to remain within clinically acceptable ranges.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for inclusion in this study must meet all of the following inclusion criteria:
* Patient ≥ 18 years old;
* Patient with confirmed CAD, with indication for elective PCI;
* Patient with CAD presenting the following specifications:

  * de novo native coronary artery lesion (i.e. a coronary lesion not previously treated)
  * Study reference vessel diameter is between 2.5 mm and 4.0 mm by visual estimate
  * Study lesion diameter showing stenosis of at least 50% by visual estimate.
* Subject deemed appropriate for robotic-assisted PCI with R-Two system used per its intended use; based on the investigator's judgment;
* The patient provides written informed consent as approved by the applicable Ethics Committee and is willing to comply with all study requirements including 30 day follow-up;
* The patient is affiliated with a social security system.
* Female subjects must be of non-child bearing potential, or if able to bear children, have a negative urinary pregnancy test within 7 days prior to the intended index procedure.

Exclusion Criteria:

* Planned PCI or coronary artery bypass graft (CABG) within 30 days after the study procedure.
* Acute myocardial infarction within 72 hours before the study procedure.
* Left ventricular ejection fraction < 30%.
* Recent PCI within 72 hours, or PCI within the past 30 days with a major adverse cardiac event.
* Known allergy or contraindication to study-related medications or materials (aspirin, heparin, P2Y12 inhibitors, stainless steel, cobalt chromium, contrast media) not manageable with premedication.
* Significant blood count abnormalities (platelets < 100,000/mm³ or > 700,000/mm³; WBC < 3,000/mm³).
* Severe renal impairment (serum creatinine > 2.0 mg/dL or eGFR < 30 mL/min).
* Stroke within 30 days before the procedure.
* Hemodynamic instability or acute pulmonary edema.
* Significant active bleeding or high bleeding risk (recent GI bleeding, bleeding disorders, refusal of transfusion).
* Pregnancy, breastfeeding, or planning pregnancy before study completion.
* Current participation in another investigational study without completed follow-up.
* Angiographic exclusions: total occlusion, intraluminal thrombus, need for atherectomy or other non-balloon devices before stenting, unprotected left main stenosis > 50%, or certain bypass graft lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Technical success | Periprocedural
  The technical success is defined as the rate of the robotic-assisted PCI completed without total manual conversion due to irretrievable technical issue or platform limitation leading to the inability of the devices to navigate vessel anatomy.

SECONDARY OUTCOMES:
Clinical success | Within 48 hours of the procedure or prior to hospital discharge, whichever occurs first
  Less than 30% of residual stenosis post PCI in the lesions treated using the robotic system without target lesion failure (TLF) either within 48 hours of the procedure or prior to hospital discharge, whichever occurs first.
Absence of intra-procedural vascular complications | Periprocedural
Absence of target lesion failure (TLF) | Hospital discharge visit 30-days follow up visit
Absence of other device-related complications | Hopistal discharge visit 30-days follow-up visit
Total and robotic procedure duration | Periprocedural
Fluoroscpoy time | Periprocedural
Radiation exposure for the patient and the primary operator | Periprocedural
  Dose of radiation exposure for the patient and the primary operator
Score of operator ergonomic assessment scale | Periprocedural
  This questionnaire is designed to assess your perceived ergonomic experience when using a robotic system compared to performing the same procedure manually. It covers several dimensions including physical, cognitive, organizational, environmental, and functional ergonomics.
Robotic precision as assessed by the rate of the longitudinal geographical miss | Procedure visit
  The longitudinal geographical miss is determined by a core lab using a quantitative coronary angiography (QCA). Longitudinal geographic miss is defined as cases where the entire length of the injured or stenotic segment was not fully covered by the total length of the stent.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre cardiologique du nord, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No